CLINICAL TRIAL: NCT05334225
Title: Assessing the Knowledge and Self-confidence of Healthcare Workers to Perform Transurethral Catheterization: A Multicenter Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Betül Kartal (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Betül Kartal, Research Coordinator/Specialist, Medipol University
Organization: Medipol University (Other)
Other Study IDs: 10010
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Urethral Catheterization; Urethral Catheterization Related Injury; Catheter Complications; Catheter Related Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Workers: Doctors, nurses, paramedics, midwifes
  Interventions: Other: Training Program

INTERVENTIONS:
Other: Training Program — An in-person urethral catheterization training program that utilizes training videos (demonstrating procedures, providing examples of ordinary and difficult cases, utilizing animation techniques as well)

SUMMARY:
Rationale: Healthcare professionals regularly perform transurethral catheterization. They may have not sufficient knowledge, experience, and self-confidence about urethral catheterization. This can cause an increased risk of urethral catheterization-related injury and morbidity. With an appropriate training program, we can raise the knowledge and self-confidence of healthcare professionals in performing transurethral catheterization.

Primary Objective: To compare knowledge and self-confidence amongst healthcare workers in performing urethral catheterization before and after the proposed urethral catheterization training program.

Secondary Objective: To compare the traumatic catheterization rates before and after the proposed urethral catheterization training program.

Study design: This study is a prospective multi-center trial using a questionnaire for assessing the healthcare professionals about urethral catheterization knowledge and self-confidence before and after a urethral catheterization training program, where their evaluation is scheduled 6 months after the training.

Study population: The study population comprises medical health workers (nurses, paramedics and doctors) from 5 different Medipol Hospitals working at surgical and non-surgical departments.

Intervention: An in-person urethral catheterization training program that utilizes training videos (demonstrating procedures, providing examples of ordinary and difficult cases, utilizing animation techniques as well) Main study parameters/endpoints: Primary endpoint is the change in self-reported self-confidence and knowledge in urethral catheterization following the training. The secondary endpoint is the change in complicated/traumatic urethral catheterization following the training. A complicated/traumatic catheterization is defined as a urethral catheterization requiring the intervention of a urologist.

ELIGIBILITY:
Inclusion Criteria: Healthcare workers (paramedics, nurses, and doctors) working in the emergency department, intensive care, operating rooms, departments of gynecology, general surgery, urology, orthopedics, neurology, internal medicine, cardiology, and anesthesiology -

Exclusion Criteria: Healthcare workers that not working non-clinic services,

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare workers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Studying The Reason For Traumatic Catheterization Through Surveys | 1 year
  Evaluating the reason why traumatic catheterization happens (lack of experience, stress, challenging case, wrong equipment, etc.) through surveys prepared for health care workers that are involved in catheterization process.
Reducing The Traumatic Catheterization Case Number Through The Training and Comparison Surveys | 1 year
  After the initial survey results, health care workers will go through a special training period for relearning correct catheterization methods. After the training, case numbers will be compared to before the training period and same survey will be distributed again to health care workers to compare their initial and final survey results.

CONTACTS AND LOCATIONS:
Overall Officials: Özgür Arıkan, Study Director — oarikan@medipol.edu.tr
Locations (1):
- Medipol Mega University Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided by request according to the primary objectives of the IPD study and according to the availability in the present trial

REFERENCES:
- [Derived] Calik G, Bahadir Z, Madendere B, Arikan O, Guzelburc V, Evci E, Cakir SS, Altay B, Laguna P, Kocak M, Albayrak S, Horuz R, Sabuncu K, Boz M, Erkurt B, Alrifaai MA, Al Chaabawi A, Alrais M, Ali IA, Ashour SMS, de la Rosette J. Knowledge and self-confidence of healthcare workers to perform transurethral catheterization: a matter deserving attention! World J Urol. 2025 May 16;43(1):311. doi: 10.1007/s00345-025-05677-3. PMID 40377708